CLINICAL TRIAL: NCT05979584
Title: Platelet Rich Plasma VS Platelet Fibrin Plasma in Treatment of Diabetes Related Wound：a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Long2023-DFU-PFP
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot
Keywords: Diabetes foot ulcer; Platelet Rich Plasma; Platelet Fibrin Plasma
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet Fibrin Plasma (Experimental): Participants of intervention group will receive Platelet Fibrin Plasma in addition with clinical optimal treatment plan after the wound bed preparation for closure.
  Interventions: Device: Platelet Fibrin Plasma
- Platelet Rich Plasma (Placebo Comparator): Participants of intervention group will receive Platelet Rich Plasma in addition with clinical optimal treatment plan after the wound bed preparation for closure.
  Interventions: Device: Platelet Rich Plasma

INTERVENTIONS:
Device: Platelet Fibrin Plasma — Participants of intervention group will receive Platelet Fibrin Plasma in addition with clinical optimal treatment plan after the wound bed preparation for closure.
  Arms: Platelet Fibrin Plasma
Device: Platelet Rich Plasma — Participants of intervention group will receive Platelet Rich Plasma in addition with clinical optimal treatment plan after the wound bed preparation for closure.
  Arms: Platelet Rich Plasma

SUMMARY:
The goal of this randomized control trial is to compare the efficacy and safety of Platelet Rich Plasma VS Platelet Fibrin Plasma in patients with diabetes foot ulcer. The main question it aims to answer are:

* Whether the Platelet Fibrin Plasma have noninferior efficacy than Platelet Rich Plasma in treatment of diabetes foot ulcer？
* Whether the Platelet Fibrin Plasma have noninferior safety than Platelet Rich Plasma in treatment of diabetes foot ulcer？ Participants will be assigned with a 1:1 ratio into intervention group and control group.

Participants of intervention group will receive Platelet Fibrin Plasma in addition with clinical optimal treatment plan after the wound bed preparation for closure. Participants of intervention group will receive Platelet Rich Plasma in addition with clinical optimal treatment plan after the wound bed preparation for closure.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is aged 18-80 years old;
2. Diagnosed as type 1 or type 2 diabetes according to the World Health Organization standard, blood sugar has been controlled before enrollment, and the level of Glycated hemoglobin HbA1c is less than 10%;
3. diabetes wounds with poor healing or prolonged healing need standard wound treatment;
4. There is no disseminated infection or the disseminated infection has been controlled;
5. After preparing the wound bed, the condition for using platelet plasma to close the wound is met;
6. Voluntarily sign an informed consent form;

Exclusion Criteria:

1. Severe diseases such as acute myocardial infarction, heart failure, hepatitis, shock, and respiratory failure have not been corrected yet;
2. Severe ischemia of the wound surface, unable to seek medical attention or not yet corrected;
3. Uncontrolled systemic or disseminated infections;
4. Blood glucose is out of control or not yet effectively controlled;
5. Blood system diseases with uncorrected coagulation dysfunction or platelet dysfunction;
6. There is active bleeding inside the wound, and routine basic treatment plans cannot be implemented;
7. Platelets ≤ 80 × 10^9, hemoglobin<90g/L;
8. Patients with advanced malignant tumors;
9. Active period of autoimmune diseases;
10. The patient is unable to cooperate or has mental disorders;
11. According to the judgment of the researchers, the patient has a clear and irremovable cause that affects wound healing, which is not suitable for this study or cannot comply with the requirements of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-09 (Actual)

PRIMARY OUTCOMES:
4-week wound healing rate | 4-week
  By D28, the proportion of healed wounds in the total number of cases

SECONDARY OUTCOMES:
The 4-week wound area reduction rate | 4-week
  (pre-treatment wound area - post-treatment wound area)/pre-treatment wound area × 100%
The 8-week wound healing rate | 8-week
  by the end of 8 weeks, the proportion of healed wounds to the total number of cases
Total blood volume required to prepare platelet plasma | day 0
Extracted platelet plasma volume | day 0
adverse events related to blood collection during the follow-up period | during the follow-up period
  such as ecchymosis/hematoma/bleeding, thrombophlebitis, and unstable circulation
Infection evaluation | during the follow-up period
  0 points for no infection and 1 point for local infection reduction, 2 points for local infection maintenance or aggravation, and 3 points for disseminated infections

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University 3rd Hospital, Beijing, Beijing Municipality, China